CLINICAL TRIAL: NCT06377839
Title: Assessment of Chronic Pain Predictors Following Surgical Removal of Mandibular Third Molars
Brief Title: Pain After Removal of Mandibular Third Molars With or Without Advanced Platelet-rich Fibrin
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Thomas Starch-Jensen, DDS, Professor, consultant surgeon, DDS, PhD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20230048
Record Dates: First submitted 2024-04-09; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Pain Syndrome
Keywords: Pain, surgery, quality of life,
MeSH Terms: conditions — Somatoform Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With advanced platelet-rich fibrin in the ekstraction socket (Active Comparator): Right or left side of the mandible
  Interventions: Biological: Advanced platelet-rich fibrin in the ekstraction socket
- Without advanced platelet-rich fibrin in the ekstraction socket (Placebo Comparator): Right or left side of the mandible
  Interventions: Biological: Advanced platelet-rich fibrin in the ekstraction socket

INTERVENTIONS:
Biological: Advanced platelet-rich fibrin in the ekstraction socket — Advanced platelet-rich fibrin is a centrifuged fibrin matrix composed of concentrated growth factors, platelet cytokines, and blood cells, which possesses the ability to stimulate wound healing and tissue regeneration. Advanced platelet-rich fibrin is manufacturing from a blood sample.

SUMMARY:
Pain is the most common complication following surgical removal of an impacted mandibular third molar. Several risk factors may increase the intensity and duration of pain following removal of mandibular third molars. Acute postoperative pain can transcript into postoperative chronic pain without an explainable reason or a specific risk factor. The use of advanced platelet-rich fibrin in the extraction socket following surgical removal of mandibular third molar have diminished the intensity and duration of acute postoperative pain and facilitated improved wound healing. The objective of the present study is therefore to identified specific risk factors and predictors for developing postoperative chronic pain following surgical removal of mandibular third molars with or without advanced platelet-rich fibrin applied in the extraction socket using epigenetic modulation.

DETAILED DESCRIPTION:
Pain is the most common complication following surgical removal of an impacted mandibular third molar (SRM3). Acute postoperative pain (APP) following SRM3 is a normal physiological response to the tissue damage and usually treated sufficiently by paracetamol, non-steroidal anti-inflammatory drugs, or opioids. Increasing age, gender, smoking habit, length of surgery, type of anesthesia, intraoperative complications, surgeon's experience, and contamination of the surgical wound are well-known risk factors that affects the intensity and duration of APP. However, APP can transcript into postoperative chronic pain (PCP) without an explainable reason or a specific risk factor. Moreover, specific predictors for development of PCP following SRM3 is currently not sufficiently elucidated.

PCP is defined as pain lasting for two months or more after surgery, when other causes of pain are excluded. The characteristics and intensity of PCP varies among individuals and specific factors for developing PCP has not yet been clearly elucidated. PCP leads to severe functional limitations and impaired oral health-related quality of life (OHRQoL). The presence of pain prior to surgery as well as the intensity and duration of APP are considered as critical predictors for developing PCP. Various pharmacological and preventive strategies have therefore been proposed to minimize the risk of APP following SRM3 including modification of the surgical technique, sufficient intra- and postoperative pain control as well as preoperative psychological intervention focusing on the psychosocial and cognitive risk factors. Moreover, risk factors, such as genetic and epigenetic modifications have also been associated with APP and PCP. Among epigenetic modifications, non-coding RNAs have shown to be associated with the development of PCP. However, clarification of factors that specifically influence the development of PCP following SRM3 remains unknown.

Advanced platelet-rich fibrin (APRF) is a centrifuged fibrin matrix composed of concentrated growth factors, platelet cytokines, and blood cells, which possesses the ability to stimulate wound healing and tissue regeneration. Manufacturing of APRF from blood samples and application of APRF in the extraction socket following SRM3 have diminished the intensity and duration of APP and facilitated improved wound healing, as reported in systematic reviews and meta-analyses. Application of APRF in the extraction socket following SRM3 possess therefore the ability to minimize the risk of developing PCP due to a shorter period of APP.

The objective of the present study is therefore to identified specific predictors for developing PCP following SRM3. Eighty patients with an impacted mandibular third molar will be randomly allocated to SRM3 with or without application of APRF in the extraction socket. A standardized postoperative pain-management regime will be applied following SRM3. Blood samples (80mL) will be obtained intraoperative and one week postoperatively for all included patients. The investigated non-coding RNAs in the blood of participants will be used to assess their association with pain sensitivity and risk of developing PCP. Self-administrated questionnaires and visual analogue scale (VAS) will be used to correlate the results of the of non-coding RNA dysregulation with the duration and intensity of postoperative pain, social and working isolation, physical appearance, eating and speaking ability, diet variations, sleep impairment, and discomfort after one week, one month, and one year, respectively. The Modified Dental Anxiety Scale is used to measure preoperatively dental anxiety. OHRQoL is evaluated by self-administrated questionnaires obtained preoperatively and compared with postoperative assessment after one week, one month, and one year. The primary outcome measure is intensity and duration of postoperative pain following SRM3 with or without application of APRF in the extraction socket. These results will be correlated with alteration in non-coding RNAs expression to identified possible predictors for developing PCP. The results will be published in international peer-reviewed journals as well as presented at congresses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Presence of a semi- or fully impacted mandibular third molar.
* Indication for surgical removal of mandibular third molar.

Exclusion Criteria:

* Patients suffering from chronic pain syndrome.
* Patients in need of daily analgetic.
* Pregnancy.
* Psychiatric problems or unrealistic expectations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of postoperative pain by using Visual Analoque scale | Postoperative (15 days)
  Measurements of pain using Visual Analogue Scale (0 is no pain and 100 is the worst pain), so lower score is a better outcome

SECONDARY OUTCOMES:
Assessment of quality of life | Pre- and postoperative (1-year)
  Questionnaire for assessment of quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial surgery, Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No